CLINICAL TRIAL: NCT00804037
Title: Injection Snoreplasty: Comparison Between Ethanol and Ethanolamine Oleate. A Randomized, Placebo-Controlled Study in Human Patients
Brief Title: Injection Snoreplasty: Comparison Between Ethanol and Ethanolamine Oleate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Fabio Lorenzetti, University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORLHCFMUSP 1
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-11

CONDITIONS: Snoring; Apnea
Keywords: Snoring and Mild Apnea
MeSH Terms: conditions — Snoring; Apnea

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ethanol (Active Comparator)
  Interventions: Procedure: Injection Snoreplasty
- Ethanolamine Oleate (Active Comparator)
  Interventions: Procedure: Injection Snoreplasty

INTERVENTIONS:
Procedure: Injection Snoreplasty — Injection of 0,5 ml of the sclerosing agent into the soft palate (3 points)

SUMMARY:
SUMMARY INTRODUCTION: among various treatments for patients with primary snoring, upper airway resistance syndrome (UARS) and obstructive sleep apnea syndrome (OSAS), the injection snoreplasty arose as a promising alternative in some selected cases.

OBJECTIVE: to investigate the efficacy and tolerance of injection snoreplasty comparing Ethanol and Ethanolamine Oleate.

ELIGIBILITY:
Inclusion Criteria:

* Snoring
* RDI < 15 /h

Exclusion Criteria:

* BMI > 35

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Snoring | 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fabio TM Lorenzetti, MD, Principal Investigator — University of Sao Paulo; Michel B Cahali, PhD, Study Director — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil